CLINICAL TRIAL: NCT04137757
Title: Neural Correlates of Cognitive Dysfunction in Postural Tachycardia Syndrome
Brief Title: fMRI in Postural Tachycardia Syndrome
Acronym: POTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Amy Arnold, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Study00012860; UL1TR002014 (NIH)
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Body Negative Pressure (LBNP) (Experimental): Participants complete mental tasks and imaging while undergoing lower body negative pressure (LBNP).
  Interventions: Other: Lower Body Negative Pressure
- Sham Pressure (Sham Comparator): Participants complete mental tasks and imaging with pressure noise but no pressure.
  Interventions: Other: Sham Pressure

INTERVENTIONS:
Other: Lower Body Negative Pressure — Lower body negative pressure will be applied.
  Arms: Lower Body Negative Pressure (LBNP)
Other: Sham Pressure — Noise will be turned on but no pressure will be applied.
  Arms: Sham Pressure

SUMMARY:
Postural tachycardia syndrome (POTS) is one of the most common forms of chronic orthostatic intolerance in the United States. This is a disabling disorder characterized by an excessive increase in heart rate upon standing that is accompanied by symptoms such as dizziness and fatigue. One of the most under appreciated and bothersome symptoms of POTS is impaired cognition or "brain fog," which occurs to a level that interferes with daily activities such as work and education. Despite this high impact, the reasons why POTS patients have problems with cognition are not well understood. This project will test the overall hypothesis that "brain fog" in POTS is related to increased activation of cognitive brain regions during mental tasks when compared with healthy subjects, and that this activation is exacerbated by in the presence of orthostatic stress.

DETAILED DESCRIPTION:
A randomized, double blind, crossover study will be conducted to determine if there are differences in resting brain structure and blood oxygen perfusion in postural tachycardia syndrome (POTS) compared with healthy subjects, and to identify the pattern of brain activation produced by cognitive testing under resting conditions and in the presence of a physical challenge mimicking orthostatic stress (lower body negative pressure, LBNP). This is an outpatient study that requires a screening visit in the Clinical Research Center within the Penn State Hershey Medical Center, and if eligible, two study visits in the Penn State Center for Nuclear Magnetic Resonance Imaging involving blood oxygen level dependent functional magnetic resonance imaging (BOLD-fMRI) and a cognitive test while lying in a magnetic resonance imaging (MRI) scanner with the lower body placed in the LBNP chamber. The LBNP chamber applies suction to the lower body to pool blood in the legs and physiologically mimic what happens when standing up. Blood pressure, heart rate, and oxygen saturation will be measured throughout the study. A scan will be performed while at rest to look at the structure and blood oxygen perfusion in the brain. The LBNP or sham pressure will then be initiated, with the order determined randomly and the other stress applied at the second study visit. Once the appropriate level of pressure is achieved, brain oxygen perfusion will be measured and subjects will be asked to complete one test of cognitive function. At the end of the cognitive test, brain oxygen levels will be measured and the testing will end. The time inside the MRI scanner at each study visit will be approximately 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races or ethnicity
* Age 18-60
* Healthy volunteers or previously diagnosed with POTS by current consensus criteria (rise in heart rate of at least 30 beats/minute within 10 minutes of standing; absence of orthostatic hypotension defined as a drop in blood pressure greater than 20/10 mmHg within 3 minutes of standing; and presence of daily orthostatic symptoms for at least 6 months such as lightheadedness, dizziness, nausea, and palpitations).
* Healthy participants must have cognitive testing scores within normal range (defined by Stroop word-color test score between 40-70) and be able to tolerate lower body negative pressure.
* POTS participants must have either mild cognitive dysfunction (defined by Stroop word-color t-score <40 and >30) or normal cognitive function (defined by Stroop word-color test score between 40-70), and able to tolerate lower body negative pressure.
* Capable of giving informed consent
* Fluent in written and spoken English

Exclusion Criteria:

* Age <18 years or >60 years
* Pregnant or breastfeeding women
* Left handedness
* Require glasses for vision correction (contact lenses are okay)
* Current smokers
* Alcohol or drug abuse
* Recreational drug use (e.g. cannabis, heroin, cocaine)
* Other potential causes for tachycardia (e.g. prolonged bed rest, dehydration)
* Taking selective norepinephrine reuptake inhibitors or stimulant medications within the past 3 months as these may alter cognition
* Unable to tolerate an MRI scanner (e.g. claustrophobia, implanted metal)
* Unable to give or withdraw informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Brain Region Activation | 60 minutes
  The change in activation of cognitive brain regions measured by blood oxygen dependent functional magnetic resonance imaging following cognitive tasks and orthostatic stress.

SECONDARY OUTCOMES:
Brain Oxygen Perfusion | 60 minutes
  The change in brain oxygen perfusion measured by arterial spin labeling magnetic resonance imaging following cognitive tasks and orthostatic stress.
Blood Pressure | 60 minutes
  The change in blood pressure following cognitive tasks and orthostatic stress.
Heart Rate | 60 minutes
  The change in heart rate following cognitive tasks and orthostatic stress.
Stroop Word-Color Score | 10 minutes
  The change in the Stroop word-color test score following orthostatic stress and sham stress. This test measure executive function. The scores are T-scores normalized to population averages based on age and education level from 0 to 100. A higher score indicates better executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Arnold, Ph.D., Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No